CLINICAL TRIAL: NCT04741490
Title: A Single-arm, Exploratory Clinical Study of Camrelizumab Combined With Radiotherapy for Adjuvant Treatment of Esophageal Squamous Cell Carcinoma After Surgery
Brief Title: Camrelizumab Combined With Radiotherapy for Adjuvant Treatment of Esophageal Squamous Cell Carcinoma After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-FJ-BC-EC-II-003
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Squamous Cell Carcinomas
MeSH Terms: interventions — camrelizumab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): The adjuvant treatment of radiotherapy combined with carrilizumab lasted for 6 cycles
  Interventions: Drug: Camrelizumab; Radiation: radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — PD-1antibodies，200mg ivgtt Q3W
Radiation: radiotherapy — 45-55Gy/1.8～2.0Gy

SUMMARY:
This is an investigator-initiated, single-arm, single-center, exploratory clinical study.The study population consisted of patients with R0 resection of esophageal squamous cell carcinoma who had not received radiation therapy.The purpose of this study was to evaluate the efficacy and safety of carrelizumab combined with radiotherapy in the adjuvant treatment of esophageal squamous cell carcinoma after surgery.About 20 subjects are planned to be enrolled in this study.Drug regimen: Patients with esophageal squamous cell carcinoma received radiotherapy combined with carrilizumab adjuvant therapy for 6 cycles 1-3 months after R0 resection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 year，male or female；
* The clinical stages of esophageal squamous cell carcinoma diagnosed by pathology (including histology or cytology) were T1-4AN0M0 and T1-4AN +M0
* Patients who underwent surgical resection and were assessed as R0.However, patients who have received previous radiotherapy should be excluded
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
* Survival expectation ≥ 3 months;
* The laboratory test value of the patient before medication should meet the following standards:

  1. Routine blood：WBC≥3.0 × 109/L；ANC≥1.5 × 109/L；PLT≥90 × 109/L；HGB≥9.0 g/dL；
  2. Liver function：TBIL≤1.5 × ULN，AST≤2.5 × ULN，ALT≤2.5 × ULN（Subjects with liver metastasis，AST≤5× ULN，ALT≤5 × ULN）；
  3. Renal function：Cr≤1.5 × ULN or CrCl ≥50 mL/min；
  4. Blood coagulation function：INR≤1.5，APTT≤1.5 ×ULN ；
* Women of childbearing age must have a serum pregnancy study within 2 weeks prior to the first dose and the results are negative. Female subjects of childbearing age and partners who are women of childbearing age must be contraceptive during the study period and within 180 days after the last administration of the study drug;

Exclusion Criteria:

* Known or suspected history of active autoimmune diseases, autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes)
* Have a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or history of organ transplantation and bone marrow transplantation；
* Interstitial lung disease, drug-induced pneumonia, radiation pneumonitis requiring steroid therapy or active pneumonia with clinical symptoms or severe pulmonary dysfunction；
* There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina (3) myocardial infarction within 24 weeks (4) clinical need for treatment or Interventional supraventricular or ventricular arrhythmia；
* Have a tendency to hereditary bleeding or coagulopathy. Clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood++ and above；
* Has not fully recovered from toxicity and/or complications from any intervention prior to initiation of treatment (i.e., ≤ grade 1 or level required at baseline, excluding fatigue or hair loss);
* Allergic reactions to test drugs for this application；
* Pregnant or lactating women；
* Those whom the investigator considered unsuitable for inclusion。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
1-year disease-free survival rate (1-year DFS) | up to approximately 1 year
  The percentage of subjects who were free of disease recurrence or death from the start of study enrolment to 12 months later.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 2 year
  the time from treatment to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.
Disease-free survival (DFS) | up to approximately 2 year
  The time from enrolment (ICF signing) to disease recurrence or death due to disease progression.
Overall survival (OS) | up to approximately 3 year
  the time between subjects' death from various causes.For subjects still alive at the last follow-up, their OS was measured as data deletion by the time of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided